CLINICAL TRIAL: NCT00528060
Title: Pilot Study to Measure Exposure to Atazanavir, as a Component of Pharmacokinetic Parameters and Adherence Measured With MEMS in Naive HIV-infected Patients Treated Once Daily With Atazanavir Combined to Ritonavir and to Tenofovir/Emtricitabine. ANRS 134 Cophar 3
Brief Title: Measure of Pharmacokinetic Parameters and Adherence With MEMS in Naive HIV Infected Patients Treated With Reyataz Once Daily Combined With Norvir and Truvada
Acronym: ANRS134COPHAR3
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Collaborators: Bristol-Myers Squibb (Industry); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-003203-12
Record Dates: First submitted 2007-09-10; First posted 2007-09-11 (Estimated); Last update posted 2011-12-22 (Estimated); Status verified 2011-12

CONDITIONS: HIV Infections
Keywords: HIV infections; atazanavir; Pharmacokinetics; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Atazanavir Sulfate; Ritonavir; Tenofovir; Emtricitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Atazanavir — 2pills/day
Drug: Ritonavir — 1 pill/day
Drug: Tenofovir/emtricitabine — 1 pill/day

SUMMARY:
the trial assessed the pharmacokinetics and long term plasma exposure of the following antiretrovirals: atazanavir when combined to ritonavir and the tenofovir/emtricitabine fixed-dose combination. All drugs will be delivered in MEMS electronic device to monitor dosing history.

DETAILED DESCRIPTION:
The trial is a phase II, open label, non-randomized, prospective multicenter trial to assess the pharmacokinetics and long term plasma exposure of the following antiretrovirals: atazanavir when combined to ritonavir and the tenofovir/emtricitabine fixed-dose combination. All drugs will be delivered in MEMS electronic device to monitor dosing history.

ELIGIBILITY:
Inclusion Criteria:

* Naïve of treatment HIV -1 infected patients
* CD4 above 100/mm3

Exclusion Criteria:

* pregnancy
* renal failure
* hepatitic disease
* ongoing opportunistic disease
* Hb under 8g/dl; platelets under 50 000/mm3; neutrophils under 750/mm3; Prothrombin index under 80%, Ca or Ph > 2.5 N
* drugs interacting with investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-01; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic parameters of atazanavir (ATV) when combined with ritonavir (RTV) and tenofovir/emtricitabine | week 4

SECONDARY OUTCOMES:
pharmacokinetics of emtricitabine and tenofovir; intraindividual variability in ARVs concentrations; adherence measured with MEMS records and validated ANRS observance autoquestionnaire; relationships between virological response or side event occurrence | Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Cécile Goujard, MD, Principal Investigator — AP-HP Kremlin-Bicetre; France Mentre, PHD, Study Director — AP-HP Bichat, Inserm U738
Locations (2):
- France (2):
  - Hopital du Kremlin Bicêtre Service de médecine interne, Kremlin Bicëtre
  - Hopital Bichat CIC, Paris

REFERENCES:
- [Derived] Parienti JJ, Barrail-Tran A, Duval X, Nembot G, Descamps D, Vigan M, Vrijens B, Panhard X, Taburet AM, Mentre F, Goujard C. Adherence profiles and therapeutic responses of treatment-naive HIV-infected patients starting boosted atazanavir-based therapy in the ANRS 134-COPHAR 3 trial. Antimicrob Agents Chemother. 2013 May;57(5):2265-71. doi: 10.1128/AAC.02605-12. Epub 2013 Mar 4. PMID 23459496